CLINICAL TRIAL: NCT07073313
Title: Using Muscle Functional MRI to Study Spatial Muscle Activation Patterns in People With SCI
Status: Not yet recruiting | Type: Observational
Sponsor: Kessler Foundation (Other)
Responsible Party: Principal Investigator, Peter Barrance, Senior Research Scientist, Kessler Foundation
Other Study IDs: R-1295-25
Record Dates: First submitted 2025-05-29; First posted 2025-07-18 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-05

CONDITIONS: Spinal Cord Injury
Keywords: Spinal Cord Injury; muscle functional MRI
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Motor incomplete Spinal Cord Injury: Chronic (>1yr) incomplete motor and sensory Spinal Cord Injury
- Able bodied control: Able bodied people with no history of lower extremity injury or gait deviation

SUMMARY:
Several types of treatment and therapy have been shown to promote improvements in movement and other health gains in people with spinal cord injury (SCI). Researchers use many different methods to measure these gains- for instance they measure their ability to stand and walk and use scanning technologies to measure bone loss and recovery. They also often use a technique known as electromyography (EMG), which detects electrical signals coming from muscles, to measure how well the muscles are being activated. While EMG has many advantages, it also has some important limitations. For instance, it is difficult to gather information from muscles below the surface, and the results can change significantly if the sensing electrodes are moved only slightly, making it harder to measure differences across different testing sessions. In this project, the investigators will use another technique to study muscle activations in people with SCI. This technique, known as muscle functional MRI (mfMRI), uses MRI scanning to measure the activation of muscles. One of the signals that MRI imaging uses has been found to change with exercise; this change is understood to be related to a buildup of chemicals in the water inside the muscle. MRI scanning has many variable settings, or parameters, that can be changed to pick up specific signals, and our team has developed a set of settings (also known as an MRI sequence) that is specially adapted to measure the mfMRI signal. Although other groups have used mfMRI to study muscle activation in other groups of people and other activities, the investigators do not believe there have been any previous studies in people with SCI. Participants in our study will lie on their back with their knee raised on a bolster and raise the lower part of their leg to straighten the knee, for several repetitions. They will do this in a room outside the MRI scanner, on a table that can be attached to the scanner for imaging. After they finish exercising, they will be moved into the MRI scan room for mfMRI scanning of the muscles of the thigh. The four muscles of the quadriceps that straighten the knee will be studied, with specialized data processing used to measure the overall activation of each of the muscles. The investigators will compare mfMRI values between people with SCI and a control group of able bodied people. These people will have motor incomplete SCI, meaning that they still have some ability to move their body in regions below the injury. By completing this study the investigators will provide new information on spatial muscle activation patterns, and they expect that this will lead the way to more widespread application of the technique in the future.

DETAILED DESCRIPTION:
Several intervention modalities including locomotor training and neuromuscular stimulation have demonstrated the ability to promote neuromuscular recovery following both motor complete and motor incomplete spinal cord injury. While an array of methodologies and technologies exist for evaluating different aspects of recovery - for instance, stabilometry to assess balance and DEXA to assess bone mineral density - there remains a need for a means to comprehensively study spatial changes to muscle activation. Electromyography (EMG) provides temporal information for muscle firing during activity; however, it has several important limitations. While surface EMG (sEMG) is relatively easily collected, it cannot collect information on deep muscles and is susceptible to cross-talk - i.e. signals originating from muscles other than those intended to be studied. Fine wire intramuscular EMG is available but is invasive, and both sEMG and fine wire EMG suffer from reliability issues related to sensitivity to exact placement of electrodes and changes in skin conductivity.

In this project the investigators propose to investigate the potential for muscle functional MRI (mfMRI) techniques to study changes in spatial patterns of neuromuscular activation associated with spinal cord injury (SCI). mfMRI imaging focuses on the time for relaxation of transverse magnetization (T2) of water in muscle, which has been found to be increased, i.e. prolonged, with exercise of the muscle. The phenomenon is understood to be related to an accumulation of osmolytes (phosphate, lactate, and sodium) in the muscle water. In our literature search the investigators have not found reports of mfMRI used to observe differences in activation in people with SCI, nor in any other neurological population. For all imaging in our study, participants will perform supine quadriceps leg raise exercises on the detachable MRI table outside the scanner. They will then be transported into the MRI scan chamber for T2 scanning of the thigh muscles. Sessions will start with several minutes of rest and baseline imaging to collect resting state T2, with exercise related T2 shifts to be calculated relative to this. Segmentation of the four quadriceps muscles on each slice will be used to describe the overall activation of each muscle. The investigators will perform a cross sectional study comparing T2 shift muscle activation values between people with motor incomplete SCI and a control group without SCI. The investigators hypothesize that people with SCI will have lower T2 shift values and less uniform muscle activation than able bodied controls. Successful completion of this study will provide new information on spatial muscle activation patterns in SCI and produce knowledge to point the way to more widespread application of the technique.

ELIGIBILITY:
Inclusion Criteria:

SCI group Inclusion criteria

* Age: 18-50 yrs
* BMI <35 kg/m2
* Chronic injury (at least 1 year post injury)
* Neurological injury status: Incomplete motor and sensory SCI classified with ASIA Impairment Scale C or D
* Ambulatory status: Participants must be nonambulatory. Individuals who can stand or walk even a few steps with or without assistance will not be eligible to participate
* Ability to flex and extend at least one knee joint under volitional control:

  * without stimulation or assistance
  * full range of motion not required
  * ability to move against gravity not required Able bodied group Inclusion criteria
* Age: 18-50 yrs
* BMI <35 kg/m2

Exclusion Criteria:

-

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: SCI group Exclusion criteria
  * Spasticity/clonus: Individuals with uncontrolled spasticity of clonus that would interfere with scanning procedures will be excluded
  * MRI contraindications including:
    * Possibility of pregnancy*
    * Implanted cardiac pacemaker
    * Cochlear implants
    * Aneurysm clip
    * Ocular metal body (e.g. metal shavings in the eye)
    * Shrapnel or bullet fragments near vital structures
    * Implanted defibrillators AB group Exclusion criteria
  * MRI contraindications including the possibility of pregnancy as listed above
  * History of injury to the dominant lower extremity
  * Any clinically significant gait deviation
  * Known factors elevating risk for stroke or heart attack during exercise
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Pattern of thigh muscle activation pattern during knee extension exercise | Baseline. The pattern will be observed one time in this single observation cross sectional study.
  T2 relaxation time values will be observed for regions of interest (ROI) for four muscles at three levels in the thigh. The T2 shift in milliseconds for each ROI will be calculated by subtracting the resting value from the value following the exercise. Hence, a T2 shift will be calculated for every muscle and imaging level. The activation pattern will be the 4x3 (muscle x level) matrix of proportions of each shift to the shifts summed across all (4x3=12) observations. In this way, the pattern represents the qualitative proportion of activation spatially across the considered muscles, and controls for differences in task performance.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Barrance, PhD, Principal Investigator — Kessler Foundation

IPD SHARING:
Plan to Share IPD: Undecided
There is no formal plan to share IPD with other researchers. The PI will cooperate with inquiries and share de-identified data and methodology details if requested.